CLINICAL TRIAL: NCT02517996
Title: Use of Preemptive Pudendal Nerve Block Prior to Hydrodistension for the Treatment of Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS): a Prospective, Double-blinded, Randomized Control Trial
Brief Title: Use of Preemptive Pudendal Nerve Block Prior to Hydrodistention for the Treatment of Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results were promising when interim analysis performed but terminated due to primary investigators left recruitment site.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00034476
Record Dates: First submitted 2015-02-23; First posted 2015-08-07 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1% Lidocaine (Experimental): Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters 1% lidocaine after anesthesia induction.
  Interventions: Drug: Lidocaine
- Normal Saline (Placebo Comparator): Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters normal saline after anesthesia induction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Total 20cc (10cc bilateral) of 1% Lidocaine: Lidocaine is a commonly used anesthetic agent suitable for infiltration, block and surface anesthesia. It is characterized by a rapid onset of action, intermediate duration of efficacy, and its elimination half-life is 90-120 minutes. Lidocaine alters signal conduction in neurons by blocking the fast voltage gated sodium (Na) channels in the neuronal cell membrane that are responsible for signal propagation. With sufficient blockage the membrane of the postsynaptic neuron will not depolarize and will thus fail to transmit an action potential. This creates the anesthetic effect by not merely preventing pain signals from propagating to the brain but by stopping them before they begin. Adverse drug reactions are rare when lidocaine is used as a local anesthetic and when administered correctly.
  Arms: 1% Lidocaine
Drug: Placebo — Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters normal saline after anesthesia induction.
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
Interstitial cystitis/Painful bladder syndrome (IC/PBS) is a chronic debilitating condition that severely impacts between 2.7 and 6.5 percent of women in the United States. Despite its public health importance the pathogenesis of IC/PBS is not well understood and there is no consensus on the optimal treatment approach for this condition. Hydrodistention is the most commonly used therapy for this condition; but it is limited by severe immediate postoperative bladder pain and its short duration of action. It has been postulated that hydrodistention works by disrupting the sensory nerves within the bladder that may be contributing to bladder pain. Recent evidence has provided support for the use of preemptive pudendal nerve block as a way to blunt immediate postoperative pain. The investigators hypothesize that preemptive pudendal nerve block prior to hydrodistention will result in lower postoperative pain after hydrodistention compared to placebo. This is a prospective double- blinded randomized study and patients will be randomized to receive preemptive bilateral pudendal nerve block with either 1% lidocaine or placebo. Bladder pain will be compared at baseline, 2 hours, 2 weeks, 6 weeks and 3 months using the Visual Analog Scale, O'Leary-Sant questionnaire and the Pelvic Pain Urgency and Frequency questionnaire.

DETAILED DESCRIPTION:
Painful bladder syndrome/interstitial cystitis (IC/PBS) is a disorder characterized by chronic bladder pain or discomfort. The exact underlying etiology of IC/PBS is unknown however several theories exist which include epithelial dysfunction, mast cell activation, and neurogenic inflammation. Whatever the underlying inciting factor for IC/PBS, the resulting phenotype is one of urinary frequency, urgency and bladder pain improved after voiding. Animal studies show that as the normal bladder fills, mechanoreceptors in the bladder wall respond to stretch through the discharge of afferent innervations or nerve firing. In normal humans, there is no conscious perception that the bladder is filling until a threshold volume is reached4. Patients with PBS/IC are thought to have substantially lower cystometric bladder volumes and a heightened sensitivity to bladder filling. Mechanoreceptors and chemoreceptors in the bladder may trigger myelinated A- delta or C-fibers found in the smooth muscle or in the submucosa in response to bladder distention. A- delta fibers are distributed mainly within the detrusor smooth muscle and are responsive to detrusor stretch that occurs during bladder filling. In contrast, C-type fibers seem to be more widespread and are distributed in the detrusor muscle, within the lamina propria and in close proximity to the urothelium. There is considerable interest in mechanisms underlying sensitization of C-fiber afferents, as these nerves are thought to play a key role in symptoms of IC/PBS. It has been shown that the plexus of afferent nerves is most dense in the regions of the bladder neck and proximal urethra. Lumbosacral afferent fibers in the pelvic and pudendal nerve, with cell bodies in the lumbosacral dorsal root ganglion (DRG), not only sense pain but also regulate continence and micturition. In laboratory animals, the pelvic nerve supply contains more stretch-responsive afferent fibers and appears to be important in responses to bladder over-distention. Neurologic changes seen after the occurrence of cystitis or other bladder insult suggest reorganization of reflex connections in the spinal cord and changes to the bladder afferents, that may suggest a greater role for the influence of the pudendal nerve on bladder pain than had been previously thought.

The pudendal nerve is a peripheral nerve that is mainly composed of afferent sensory fibers from sacral nerve roots S1, S2, and S3 and consequently it is a major contributor to bladder afferent regulation and bladder function. Pudendal nerve entrapment often leads to significant voiding dysfunction including urinary incontinence and over active bladder syndrome Furthermore, because the pudendal nerve carries such a large percentage of afferent fibers, it has been an attractive target for neuromodulation in treating refractory overactive bladder and may be useful for modulating pain experienced in IC/PBS.

No treatment has been consistently shown to provide relief in the majority of patients with painful bladder syndrome. Furthermore, combination treatment modalities are needed in the majority of patients. Cystoscopy with hydrodistention is thought to be a useful therapeutic tool in patients who are unresponsive to therapies like medication and pelvic floor physical therapy; however, its use has only been studied in a few observational studies and is currently listed as a third line treatment option for IC/PBS. According to the interstitial cystitis database study experience cystoscopy with hydrodistention is reported to be the most commonly used treatment modality for IC/PBS and published studies have reported improvement in symptoms in 70 to 80 percent of patients while other studies have reported improvement in only 40 percent. It has been postulated that hydrodistention works by disrupting the sensory nerves within the bladder that may be contributing to bladder pain and enabling the regeneration of afferent sensory nerves. Though the exact mechanism of action is unclear, there is ample evidence to suggest the efficacy of cystoscopy with hydrodistention, in a recent study by Chien-Ying et al, therapeutic hydrodistension was associated with an increase in bladder capacity and significant reduction in average O'Leary- Sant symptom and problem scores after treatment. In addition, Aihara et al who determined a positive therapeutic outcome in 71% of patients 1 month after hydrodistention have reported similar findings. The disadvantages of hydrodistention are that some patients experience a temporary worsening of their symptoms immediately following the procedure and any beneficial effect often lasts between 2-6 weeks. The immediate worsening of bladder symptoms immediately after hydrodistention and its relatively short duration of effect are often deterrents to recommending this therapy to patients. Given the multimodal approach to managing patients with IC/PBS it is imperative that the investigators explore ways to prolong the efficacy of available options and one approach that has been recently suggested is the use of preemptive analgesia.

In 1983, Woolf proposed that persistent pain experienced after trauma or surgery is due to posttraumatic functional changes not only in the peripheral pain receptors but also in the dorsal horn of the spinal cord a property known as hyperexcitability. The hyperexcitable state persists long after such stimuli cease, causing the patient to perceive pain from stimuli normally believed to be painless a common occurrence thought to be seen in patients with IC/PBS. Therefore, prevention of spinal hyperexcitability by blockade of the afferent nerve pathway from surgical site to spinal cord may therefore decrease the amount and duration of postoperative pain perception. This theory has been tested in various animal studies and was first described by Wall in 1988. In addition, the current literature on preemptive analgesia in gynecology is supportive of this approach. In a study by Ismail et al, 130 patients undergoing posterior colporrhaphy were randomized to receive preemptive pudendal nerve block with either .25% bupivacaine or normal saline. Study findings demonstrated an average postoperative Visual Analog Scale (VAS) score of 51.1 for the bupivacaine group compared to 23.5 in the placebo group. The investigators postulate that since the pudendal nerve is an important contributor to bladder afferent regulation, preemptive nerve block prior to hydrodistention may block afferent impulse transmission to the spinal cord and decrease the initial increase in postoperative bladder pain.

ELIGIBILITY:
Inclusion Criteria:

* All women aged greater than 18 years of age scheduled to undergo cystoscopy with hydrodistention
* who are literate,
* English speaking and
* can provide written informed consent will be included in this study.

Exclusion Criteria:

* Patients who have intolerance or known allergies to local analgesia will be excluded.
* In addition, patients who have coagulation disorders will also be excluded as this may increase their risks of complication from bleeding.
* Patient will also be excluded if they have a history of dementia as this may impair their ability to follow instructions.
* Patients who are non-ambulatory and who have an inability to fully assess pain will also be excluded.
* Patients receiving additional surgical procedures will be excluded from the study, as the source of their pain may be difficult to decipher in the immediate post-operative period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tola Fashokun, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] De Groat WC. Nervous control of the urinary bladder of the cat. Brain Res. 1975 Apr 11;87(2-3):201-11. doi: 10.1016/0006-8993(75)90417-5. No abstract available. PMID 1125771
- [Background] GARRY RC, ROBERTS TD, TODD JK. Reflexes involving the external urethral sphincter in the cat. J Physiol. 1959 Dec;149(3):653-65. doi: 10.1113/jphysiol.1959.sp006366. No abstract available. PMID 13826682
- [Background] Birder L, de Groat W, Mills I, Morrison J, Thor K, Drake M. Neural control of the lower urinary tract: peripheral and spinal mechanisms. Neurourol Urodyn. 2010;29(1):128-39. doi: 10.1002/nau.20837. PMID 20025024
- [Background] Kuo YC, Kuo HC. The urodynamic characteristics and prognostic factors of patients with interstitial cystitis/bladder pain syndrome. Int J Clin Pract. 2013 Sep;67(9):863-9. doi: 10.1111/ijcp.12116. PMID 23952465
- [Background] Malykhina AP. Neural mechanisms of pelvic organ cross-sensitization. Neuroscience. 2007 Nov 9;149(3):660-72. doi: 10.1016/j.neuroscience.2007.07.053. Epub 2007 Sep 8. PMID 17920206
- [Background] Pezzone MA, Liang R, Fraser MO. A model of neural cross-talk and irritation in the pelvis: implications for the overlap of chronic pelvic pain disorders. Gastroenterology. 2005 Jun;128(7):1953-64. doi: 10.1053/j.gastro.2005.03.008. PMID 15940629
- [Background] Bruns TM, Weber DJ, Gaunt RA. Microstimulation of afferents in the sacral dorsal root ganglia can evoke reflex bladder activity. Neurourol Urodyn. 2015 Jan;34(1):65-71. doi: 10.1002/nau.22514. Epub 2014 Jan 24. PMID 24464833
- [Background] Tai C, Wang J, Wang X, de Groat WC, Roppolo JR. Bladder inhibition or voiding induced by pudendal nerve stimulation in chronic spinal cord injured cats. Neurourol Urodyn. 2007;26(4):570-577. doi: 10.1002/nau.20374. PMID 17304521
- [Background] McGee MJ, Grill WM. Selective co-stimulation of pudendal afferents enhances bladder activation and improves voiding efficiency. Neurourol Urodyn. 2014 Nov;33(8):1272-8. doi: 10.1002/nau.22474. Epub 2013 Aug 9. PMID 23934615
- [Background] Possover M, Forman A. Voiding Dysfunction Associated with Pudendal Nerve Entrapment. Curr Bladder Dysfunct Rep. 2012 Dec;7(4):281-285. doi: 10.1007/s11884-012-0156-5. Epub 2012 Sep 28. PMID 23162676
- [Background] Peters KM, Killinger KA, Boguslawski BM, Boura JA. Chronic pudendal neuromodulation: expanding available treatment options for refractory urologic symptoms. Neurourol Urodyn. 2010 Sep;29(7):1267-71. doi: 10.1002/nau.20823. PMID 19787710
- [Background] Wang S, Zhang S, Zhao L. Long-term efficacy of electrical pudendal nerve stimulation for urgency-frequency syndrome in women. Int Urogynecol J. 2014 Mar;25(3):397-402. doi: 10.1007/s00192-013-2223-7. Epub 2013 Oct 3. PMID 24091564
- [Background] Rovner E, Propert KJ, Brensinger C, Wein AJ, Foy M, Kirkemo A, Landis JR, Kusek JW, Nyberg LM. Treatments used in women with interstitial cystitis: the interstitial cystitis data base (ICDB) study experience. The Interstitial Cystitis Data Base Study Group. Urology. 2000 Dec 20;56(6):940-5. doi: 10.1016/s0090-4295(00)00845-1. PMID 11113737
- [Background] Ottem DP, Teichman JM. What is the value of cystoscopy with hydrodistension for interstitial cystitis? Urology. 2005 Sep;66(3):494-9. doi: 10.1016/j.urology.2005.04.011. PMID 16140064
- [Background] Wu, C. Y., Chen, I., & Tong, Y. C. (2013). Long-term treatment outcomes in patients with interstitial cystitis/painful bladder syndrome: 10-year experience in NCKUH. Urological Science, 24(1), 10-13
- [Background] Aihara K, Hirayama A, Tanaka N, Fujimoto K, Yoshida K, Hirao Y. Hydrodistension under local anesthesia for patients with suspected painful bladder syndrome/interstitial cystitis: safety, diagnostic potential and therapeutic efficacy. Int J Urol. 2009 Dec;16(12):947-52. doi: 10.1111/j.1442-2042.2009.02396.x. PMID 19817916
- [Background] Davis NF, Brady CM, Creagh T. Interstitial cystitis/painful bladder syndrome: epidemiology, pathophysiology and evidence-based treatment options. Eur J Obstet Gynecol Reprod Biol. 2014 Apr;175:30-7. doi: 10.1016/j.ejogrb.2013.12.041. Epub 2014 Jan 13. PMID 24480114
- [Background] Hsieh CH, Chang ST, Hsieh CJ, Hsu CS, Kuo TC, Chang HC, Lin YH. Treatment of interstitial cystitis with hydrodistention and bladder training. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Oct;19(10):1379-84. doi: 10.1007/s00192-008-0640-9. Epub 2008 May 22. PMID 18496634
- [Background] Yamada T, Murayama T, Andoh M. Adjuvant hydrodistension under epidural anesthesia for interstitial cystitis. Int J Urol. 2003 Sep;10(9):463-8; discussion 469. doi: 10.1046/j.1442-2042.2003.00664.x. PMID 12941123
- [Background] Cole EE, Scarpero HM, Dmochowski RR. Are patient symptoms predictive of the diagnostic and/or therapeutic value of hydrodistention? Neurourol Urodyn. 2005;24(7):638-42. doi: 10.1002/nau.20200. PMID 16208660
- [Background] Erickson DR, Kunselman AR, Bentley CM, Peters KM, Rovner ES, Demers LM, Wheeler MA, Keay SK. Changes in urine markers and symptoms after bladder distention for interstitial cystitis. J Urol. 2007 Feb;177(2):556-60. doi: 10.1016/j.juro.2006.09.029. PMID 17222633
- [Background] Woolf CJ. Evidence for a central component of post-injury pain hypersensitivity. Nature. 1983 Dec 15-21;306(5944):686-8. doi: 10.1038/306686a0. PMID 6656869
- [Background] Ke RW, Portera SG, Bagous W, Lincoln SR. A randomized, double-blinded trial of preemptive analgesia in laparoscopy. Obstet Gynecol. 1998 Dec;92(6):972-5. doi: 10.1016/s0029-7844(98)00303-2. PMID 9840560
- [Background] Ismail MT, Elshmaa NS. Pre-emptive analgesia by nerve stimulator guided pudendal nerve block for posterior colpoperineorrhaphy. Eur J Obstet Gynecol Reprod Biol. 2012 Aug;163(2):200-3. doi: 10.1016/j.ejogrb.2012.03.032. Epub 2012 Apr 27. PMID 22542612
- [Background] Long JB, Eiland RJ, Hentz JG, Mergens PA, Magtibay PM, Kho RM, Magrina JF, Cornella JL. Randomized trial of preemptive local analgesia in vaginal surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):5-10. doi: 10.1007/s00192-008-0716-6. Epub 2008 Oct 2. PMID 18830553
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Background] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Brewer ME, White WM, Klein FA, Klein LM, Waters WB. Validity of Pelvic Pain, Urgency, and Frequency questionnaire in patients with interstitial cystitis/painful bladder syndrome. Urology. 2007 Oct;70(4):646-9. doi: 10.1016/j.urology.2007.06.1089. Epub 2007 Aug 20. PMID 17707887
- [Background] Parsons CL, Dell J, Stanford EJ, Bullen M, Kahn BS, Waxell T, Koziol JA. Increased prevalence of interstitial cystitis: previously unrecognized urologic and gynecologic cases identified using a new symptom questionnaire and intravesical potassium sensitivity. Urology. 2002 Oct;60(4):573-8. doi: 10.1016/s0090-4295(02)01829-0. PMID 12385909
- [Background] Lowenstein L, Zimmer EZ, Deutsch M, Paz Y, Yaniv D, Jakobi P. Preoperative analgesia with local lidocaine infiltration for abdominal hysterectomy pain management. Eur J Obstet Gynecol Reprod Biol. 2008 Feb;136(2):239-42. doi: 10.1016/j.ejogrb.2006.11.008. Epub 2006 Dec 18. PMID 17178187
- [Background] O'Neal MG, Beste T, Shackelford DP. Utility of preemptive local analgesia in vaginal hysterectomy. Am J Obstet Gynecol. 2003 Dec;189(6):1539-41; discussion 1541-2. doi: 10.1016/j.ajog.2003.10.691. PMID 14710057
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Katz J, McCartney CJ. Current status of preemptive analgesia. Curr Opin Anaesthesiol. 2002 Aug;15(4):435-41. doi: 10.1097/00001503-200208000-00005. PMID 17019235
- [Background] Pogatzki-Zahn EM, Zahn PK. From preemptive to preventive analgesia. Curr Opin Anaesthesiol. 2006 Oct;19(5):551-5. doi: 10.1097/01.aco.0000245283.45529.f9. PMID 16960490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for this study are recruited either directly from the clinic of a Urogyn attending, or are identified the week before surgery on the OR schedule. The patients eligible for this study need to be posted for cystoscopy with hydrodistention for a diagnosis of bladder pain.
Pre-assignment Details: 1 woman was unmasked after her initial postoperative scores were collected because of postoperative symptoms.
Groups:
- 1% Lidocaine: Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters 1% lidocaine after anesthesia induction.
  Lidocaine: Total 20cc (10cc bilateral) of 1% Lidocaine: Lidocaine is a commonly used anesthetic agent suitable for infiltration, block and surface anesthesia. It is characterized by a rapid onset of action, intermediate duration of efficacy, and its elimination half-life is 90-120 minutes. Lidocaine alters signal conduction in neurons by blocking the fast voltage gated sodium (Na) channels in the neuronal cell membrane that are responsible for signal propagation. With sufficient blockage the postsynaptic neuron membrane will not depolarize and so fail to transmit an action potential. This creates the anesthetic effect by not merely preventing pain signals from propagating to the brain but by stopping them before they begin. Adverse drug reactions are rare when lidocaine is used as a local anesthetic and when administered correctly.
Period: Overall Study
Arm/Group | 1% Lidocaine | Normal Saline
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Lidocaine | Normal Saline | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.1 [20 to 65] | 39.7 [29 to 55] | 40.4 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
Previous procedure [Count of Participants; unit: Participants] — Whether a patient had a previous hydrodistention procedure. Collected via a demographics form administered with all other baseline measures.
  Participants | 5 | 4 | 9
Number of other therapies [Median (Full Range); unit: Number of other therapies] — Other previous therapies for pelvic pain/pelvic floor disorders. Collected via demographic information form administered during baseline survey. Previous therapies include: pelvic floor physical therapy, bladder installations, medications, Botox injection, surgery, or herbal therapy.
  Number of other therapies | 3 [1 to 11] | 3 [1 to 9] | 3 [1 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level as Assessed by the Visual Analog Scale (VAS)
Description: To determine the change in pain at 2 hours, 2 weeks, 6 weeks, and 3 months postoperatively in patients undergoing hydrodistention with preemptive pudendal nerve block (1% Lidocaine) compared to hydrodistention with placebo (saline) using the visual analog scale (VAS).
  VAS consists of a 10cm horizontal line with the minimum endpoint labeled "no pain" (0) and maximum labeled "worst pain ever" (10). Patients placed a mark on the point that corresponds to the level of pain severity they felt. The cm distance from the low end of the VAS to the patient's mark is used as the numerical index of the intensity of pain. Pain scores of 3.0-5.4 cm are moderate, over 5.4 indicates severe pain.
Time Frame: Baseline, 2 hours, 2 weeks, 6 weeks, 3 months (Up to 3 months)
Population: Loss to follow up of 2 participants in the Normal Saline group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 1% Lidocaine: Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters 1% lidocaine after anesthesia induction.
  Lidocaine: Total 20cc (10cc bilateral) of 1% Lidocaine: Lidocaine is a commonly used anesthetic agent suitable for infiltration, block and surface anesthesia. It is characterized by a rapid onset of action, intermediate duration of efficacy, and its elimination half-life is 90-120 minutes. Lidocaine alters signal conduction in neurons by blocking the fast voltage gated sodium (Na) channels in the neuronal cell membrane that are responsible for signal propagation. With sufficient blockage the membrane of the postsynaptic neuron will not depolarize and will thus fail to transmit an action potential. This creates the anesthetic effect by stopping pain signals from propagating to the brain before they begin. Adverse drug reactions are rare when lidocaine is used as a local anesthetic and when administered correctly.
Arm/Group | 1% Lidocaine | Normal Saline
Number analyzed (Participants) | 8 | 9
score on a scale
  Pre operative VAS score: number analyzed (Participants) | 8 | 7
  Pre operative VAS score | 3.125 (2.59) | 4.5 (2.5)
  Post operative VAS score: number analyzed (Participants) | 8 | 7
  Post operative VAS score | 3.75 (2.43) | 5 (1.73)
  2 week post operative VAS scores: number analyzed (Participants) | 7 | 7
  2 week post operative VAS scores | 2.7 (2.68) | 4.8 (1.30)
  6 week post operative VAS score: number analyzed (Participants) | 5 | 3
  6 week post operative VAS score | 3 (3.31) | 4.33 (2.1)
  12 weeks post operative VAS score: number analyzed (Participants) | 5 | 2
  12 weeks post operative VAS score | 2.6 (2.4) | 2 (2.82)

2. Primary Outcome: Change in IC Symptom Index Questionnaire With Preemptive Pudendal Nerve Block Compared to Saline
Description: To determine the change in interstitial cystitis symptom index at baseline, 2 hours, 2 weeks, 6 weeks and 3 months after hydrodistention with preemptive pudendal nerve block (1% Lidocaine) compared to hydrodistention with placebo (saline).
  The IC symptom index questionnaire consists of 4 questions on IC symptoms. 2 of the questions have 6 answer choices ranging from 0-never, to 5-almost always. 1 question has 6 answer choices ranging from 0-never to 5-usually. 1 question has 7 answer choices ranging from 0-never to 6-5 or more times. The numerical score for each question are added together, with a minimum score of 0 and a maximum score of 21. A higher score indicates greater severity of IC symptoms.
Time Frame: Baseline, 2 weeks, 6 weeks, 3 months (Up to 3 months)
Population: Loss to follow up of 2 participants in the Normal Saline group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Lidocaine | Normal Saline
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline: number analyzed (Participants) | 8 | 7
  Baseline | 12.5 (3.74) | 10 (2.52)
  2 weeks: number analyzed (Participants) | 7 | 5
  2 weeks | 11.43 (4.72) | 9 (3.16)
  6 weeks: number analyzed (Participants) | 5 | 3
  6 weeks | 11.8 (3.83) | 8.67 (4.62)
  12 weeks: number analyzed (Participants) | 5 | 2
  12 weeks | 10 (3.94) | 5 (1.41)

3. Primary Outcome: Change in Problem Index (O'Leary Sant) With Preemptive Pudendal Nerve Block Compared to Saline
Description: To determine the change in problem index (O'Leary Sant) at baseline, 2 hours, 2 weeks, 6 weeks and 3 months after hydrodistention with preemptive pudendal nerve block (1% Lidocaine) compared to hydrodistention with placebo (saline).
  The IC problem index questionnaire consists of 4 questions on how much of a problem a patient's IC symptoms cause them. Each question has 5 answer choices ranging from 0-no problem, to 4-big problem. The numerical score for each question are added together, with a minimum score of 0 and a maximum score of 16. A higher score indicates that IC symptoms cause more problems for the patient.
Time Frame: Baseline, 2 hours, 2 weeks, 6 weeks, 3 months (Up to 3 months)
Population: Loss to follow up of 2 participants in the Normal Saline group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Lidocaine | Normal Saline
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline: number analyzed (Participants) | 8 | 7
  Baseline | 11.75 (2.92) | 9.43 (3.10)
  2 weeks: number analyzed (Participants) | 7 | 5
  2 weeks | 9.71 (3.95) | 8.6 (2.07)
  6 weeks: number analyzed (Participants) | 5 | 3
  6 weeks | 10 (3.81) | 7.33 (3.21)
  12 weeks: number analyzed (Participants) | 5 | 2
  12 weeks | 9.6 (2.79) | 6 (2.83)

4. Primary Outcome: Change in Pelvic Urgency, Pain, and Frequency (PUF) Questionnaire With Preemptive Pudendal Nerve Block Compared to Saline
Description: To determine the change in pelvic urgency, pain and frequency (PUF) questionnaire at baseline, 2 hours, 2 weeks, 6 weeks and 3 months after hydrodistention with preemptive pudendal nerve block (1% Lidocaine) compared to hydrodistention with placebo (saline).
  The Pelvic Urgency, Pain, and Frequency Patient Symptom Scale asks 11 questions, 7 on PUF symptoms, 4 on how bothersome PUF symptoms are. Symptom questions include 3, 4, or 5 ranked answers, with higher answers indicating more voids, or greater frequency of pain. The bother questions each of 4 ranked answers from 0-never, to 3-always. The symptom score is added, the bother score is added, and then the total score is added. The total PUF score is then reported. The minimum score is 0 and the maximum score is 35, and a higher score indicates greater symptoms and higher bother from pelvic pain and frequency.
Time Frame: Baseline, 2 hours, 2 weeks, 6 weeks, 3 months (Up to 3 months)
Population: Loss to follow up of 3 participants in the Normal Saline group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1% Lidocaine | Normal Saline
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline: number analyzed (Participants) | 8 | 6
  Baseline | 22.63 (6.74) | 19 (4)
  2 weeks: number analyzed (Participants) | 6 | 5
  2 weeks | 18.83 (7.99) | 17.4 (4.72)
  6 weeks: number analyzed (Participants) | 5 | 3
  6 weeks | 18.2 (7.53) | 16.7 (3.21)
  12 weeks: number analyzed (Participants) | 5 | 1
  12 weeks | 17.2 (6.61) | 14 (NA) — 1 participant

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data was collected from the time of the procedure to 3 months after the procedure.
Groups:
- 1% Lidocaine: Patients randomized in this arm will receive preemptive bilateral pudendal nerve block with 20 cubic centimeters 1% lidocaine after anesthesia induction.
  Lidocaine: Total 20cc (10cc bilateral) of 1% Lidocaine: Lidocaine is a commonly used anesthetic agent suitable for infiltration, block and surface anesthesia. It is characterized by a rapid onset of action, intermediate duration of efficacy, and its elimination half-life is 90-120 minutes. Lidocaine alters signal conduction in neurons by blocking the fast voltage gated sodium (Na) channels in the neuronal cell membrane that are responsible for signal propagation. With sufficient blockage the membrane of the postsynaptic neuron will not depolarize and will thus fail to transmit an action potential. This creates the anesthetic effect by preventing pain signals before they begin. Adverse drug reactions are rare when lidocaine is used as a local anesthetic and when administered.
Arm/Group | 1% Lidocaine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
Many potential participants noted that they were unwilling to enroll due to fear of being randomized to the saline arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT02517996/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02517996/ICF_001.pdf